CLINICAL TRIAL: NCT00496431
Title: Phase II Study of the Histone-deacetylase Inhibitor ITF2357 in Very High-risk Relapsed/Refractory Hodgkin's Lymphoma Patients
Brief Title: phII Study of an HDAC Inhibitor in Very High-risk Relapsed/Refractory Hodgkin's Lymphoma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study accrual was stopped earlier than planned by the Sponsor for 2 main reasons: very slow recruitment rate; lower than estimated efficacy of the drug when delivered as single agent.
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/07/2357/26; 2007-000049-36 (EudraCT Number)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — givinostat hydrochloride; givinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ITF2357 (Experimental): Patients were provided with the appropriate number of 50 mg hard gelatine capsules for oral administration for 7 days treatment, i.e. at the daily dose of 100 mg, 14 capsules 50 mg each, plus 2 spare capsules suitable in case of accidental loss.
  Interventions: Drug: histone deacetylase inhibitor (ITF2357)

INTERVENTIONS:
Drug: histone deacetylase inhibitor (ITF2357) — 50 mg b.i.d. (or every 8 hours or every 6 hours), every day
  Other Names: Givinostat

SUMMARY:
PRIMARY OBJECTIVE

- To evaluate the efficacy (according to the International Working Group response criteria for Hodgkin's Lymphomas [7, 8, 9]) of daily oral doses of ITF2357 administered to very high-risk Hodgkin's lymphoma patients.

SECONDARY OBJECTIVES

* To evaluate safety and tolerability of multiple oral doses of ITF2357
* To assess the proportion of patients that, after ITF2357 treatment, can undergo high-dose salvage chemotherapy with either autografting or allografting

DETAILED DESCRIPTION:
This is a multi-center, open label, phase II study testing ITF2357 in a population of very high-risk relapsed/refractory Hodgkin's lymphoma patients.

The patients were planned to receive 50 mg ITF2357 four times a day at 6-hour intervals in fed conditions for 28 consecutive days unless evidence of progressive disease, presence of unacceptable adverse events or patient's request to discontinue treatment occurs.

Decision regarding the continuation of ITF2357 were made on:

* the basis of tumor reassessment upon completion of cycle defined as above and not later than 7 days and
* the occurred toxicity (if any).

If complete response or partial response or stabilization of disease after first cycle, without concomitant relevant toxicities is observed, the treatment may continue as long as there is no evidence of progressive disease or appearance of unacceptable adverse events.

In any case, the treatment is not planned to exceed 84 days of drug intake overall (i.e. 12 weeks).

The treatment is planned to be administered on an outpatient basis and patients are planned to be followed regularly with physical and laboratory tests, as specified in the protocol; in case of hospitalization, the treatment will be continued or interrupted according to the Investigators' decision.

The study planned to accrue 23 patients evaluable for efficacy and the anticipated duration of the study is about 18 months.

Actually, accrual was stopped earlier than planned by the Sponsor for 2 main reasons: a) a very slow recruitment rate; b) an unplanned interim analysis suggesting a lower than estimated efficacy of the drug when delivered as single agent.

ELIGIBILITY:
Inclusion Criteria:

Signed Informed Consent Form; Age ≥ 18 years; History of histologically confirmed Hodgkin's lymphoma Subjects are eligible for this trial if (1) they have failed at least 1 cycle of chemotherapy, with or without radiotherapy, and if (2) they are considered incurable by the referring physician, and would be treated with second-line or subsequent-line salvage regimens, mainly with palliative intent; Clinical laboratory values ANC > 1500/µL; Platelet count > 75000/µL Hemoglobin > 9 g/dL (may not be transfused or treated with erythropoietin to maintain or exceed this level) Total bilirubin < 1.6 mg/dL; AST or ALT < 2.5 times the upper limit of normal Serum creatinine < 2.0 mg/dL or creatinine clearance > 50 mL/min Serum Potassium and Magnesium within normal limits; Measurable disease (according to the International Working Group response criteria for HL); ECOG performance status of 0 or 1; Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential (use per institutional standard); Life expectancy of > 3 months;; At least 4 weeks since last treatment for HL Willingness and capability to comply with the requirements of the study;

Exclusion Criteria:

Active bacterial or mycotic infection requiring antimicrobial treatment on Day 1; Pregnancy or lactation; A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval > 450 ms, according to Bazett's correction formula); The use of concomitant medications that prolong the QT/QTc interval;

Clinically significant cardiovascular disease e.g.:

Uncontrolled hypertension, myocardial infarction, unstable angina New York Heart Association (NYHA) Grade II or greater congestive heart failure History of any cardiac arrhythmia requiring medication (irrespective of its severity) Grade II or greater peripheral vascular disease A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome); Positive blood test for HIV, HBV and HCV; Identification of viral DNA by quantitative PCR for EBV (Ebstein Barr virus), JC virus, CMV (Cytomegalovirus) and Herpes Zoster; History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Total number of Objective Responses (OR): Complete Responses (CR) and Partial Responses (PR) | every 28 days
  The objective response of the patients was assessed as complete response or partial response after ITF2357 treatment.

SECONDARY OUTCOMES:
Number of subjects experiencing an Adverse Events | Throughout the study till follow-up after 3 months
  Type, frequency, severity, timing and relatedness of AEs (including changes in vital signs and clinical laboratory results) proportion of patients that, after ITF2357 treatment, can undergo high-dose salvage chemotherapy with either autografting or allografting.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Massimo Gianni, MD, Principal Investigator — Istituto Nazionale per lo studio e la cura dei Tumori (Milan - Italy)
Locations (1):
- Istituto Nazionale per lo studio e la cura dei Tumori, Milan, Italy